CLINICAL TRIAL: NCT02573389
Title: A Pilot Study on the Effect of Transampullary Pancreatic Duct Stenting on Postoperative Pancreatic Fistula Rate After Distal Pancreatectomy
Brief Title: Pancreatic Duct Stenting to Prevent Postoperative Pancreatic Fistula (POPF) After Distal Pancreatectomy
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of accrual due to competing study
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KPSC IRB 10705; KPSC IRB10705 (Other: Kaiser Permanente Southern California IRB)
Record Dates: First submitted 2015-10-07; First posted 2015-10-09 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Pancreatitis
Keywords: pancreatic fistula, pancreatectomy, endoscopic stenting, pancreatic stenting, distal pancreatectomy
MeSH Terms: conditions — Pancreatitis; Pancreatic Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Retrospective and prospective "non-stented" (No Intervention): Non-stented patients undergoing distal pancreatectomy retrospectively (2008-2015) and prospectively from 2015 to 2017.
- Prospective "stented" (Experimental): Patients who undergo prophylactic pancreatic duct stenting prior to a distal pancreatectomy starting approximately September 2015.
  Interventions: Device: Boston Scientific or Cook pancreatic duct stents

INTERVENTIONS:
Device: Boston Scientific or Cook pancreatic duct stents — Boston Scientific or Cook straight or pigtail pancreatic stents. Stent size depends on duct size (capacity). Pancreatic plastic stents are made primarily of polyethylene materials. Pancreatic stent sizes range from 2 to 25 cm in length and 3F to 11.5F in.
  Arms: Prospective "stented"

SUMMARY:
To determine whether pre-operative pancreatic stenting for distal pancreatectomy will impact the incidence of a post-operative pancreatic fistula, as defined by postoperative. If pre-operative pancreatic stenting appears to reduce the formation of Postoperative Pancreatic Fistula (POPF) in this pilot study, this will form the basis of a larger randomized trial in the future. The hypothesis is that pre-operative pancreatic duct stenting can significantly decrease the rate of development of a post-operative pancreatic fistula after distal pancreatectomy.

DETAILED DESCRIPTION:
Prophylactic pancreatic duct stenting is to be offered to all patients deemed a candidate for a distal pancreatectomy. This is a nonrandomized cohort study with a retrospective and prospective control group (Jan 2008 - Dec 2017 or sample size obtained) and a prospective endoscopic intervention group (September 2015 - Dec 2017 or until sample size obtained). We will then compare the rate of development of a postoperative pancreatic fistula between those patients who have preoperative stenting and those who do not. POPF will be defined as the amylase level of drain contents equaling three times or more the serum amylase on postoperative day 3, as defined by the International Study Group for Pancreatic Fistula (ISGPF) or an ICD-9 diagnosis of 577.8. The patient will have a pre-operative visit for stent placement and a post-operative visit for stent removal if still in place 4-6 weeks after distal pancreatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients age 18 years of age and older
2. Patients undergoing distal pancreatectomy for primary pancreatic disorder or isolated metastases to the pancreas.

Exclusion Criteria:

1. Pediatric patients younger than age 18
2. Pregnant patients
3. Patients undergoing distal pancreatectomies performed en bloc for non- pancreatic pathologies (gastric cancer, renal cell cancer, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-12-04 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative pancreatic fistula | At 6 months when enrollment begins
  Rate of post-operative pancreatic fistula will be evaluated at 6 months when enrollment begins. Early stop is determined under either of below conditions:
  * Effect size is smaller than needed to reach statistical difference even if number of enrollment is completed in one year.
  * Adverse events occurring from the pancreatic duct stenting itself, which include pseudocyst, delaying surgery, pancreatitis requiring prolonged hospital admission, or death.
  * There is statistical significant difference between control and intervention groups.

SECONDARY OUTCOMES:
Pre-operative: Pancreatitis from pancreatic duct stent | 1 - 2 weeks prior to distal pancreatectomy
Postoperative: Abscess, hemorrhage, reoperation, pulmonary embolism, mortality | 3 days post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Louis A DiFronzo, MD, Principal Investigator — Kaiser Permanente

REFERENCES:
- [Background] Jin T, Altaf K, Xiong JJ, Huang W, Javed MA, Mai G, Liu XB, Hu WM, Xia Q. A systematic review and meta-analysis of studies comparing laparoscopic and open distal pancreatectomy. HPB (Oxford). 2012 Nov;14(11):711-24. doi: 10.1111/j.1477-2574.2012.00531.x. Epub 2012 Aug 7. PMID 23043660
- [Background] Schoellhammer HF, Fong Y, Gagandeep S. Techniques for prevention of pancreatic leak after pancreatectomy. Hepatobiliary Surg Nutr. 2014 Oct;3(5):276-87. doi: 10.3978/j.issn.2304-3881.2014.08.08. PMID 25392839
- [Background] 3. American Society for Gastrointestinal Endoscopy (ASGE) Technology Assessment Committee. Status evaluation reports: Pancreatic and biliary stents. Gastrointest Endosc. 2013;77(3):319-327.
- [Background] Reddymasu SC, Pakseresht K, Moloney B, Alsop B, Oropezia-Vail M, Olyaee M. Incidence of pancreatic fistula after distal pancreatectomy and efficacy of endoscopic therapy for its management: results from a tertiary care center. Case Rep Gastroenterol. 2013 Aug 16;7(2):332-9. doi: 10.1159/000354136. eCollection 2013. PMID 24019766
- [Background] Rieder B, Krampulz D, Adolf J, Pfeiffer A. Endoscopic pancreatic sphincterotomy and stenting for preoperative prophylaxis of pancreatic fistula after distal pancreatectomy. Gastrointest Endosc. 2010 Sep;72(3):536-42. doi: 10.1016/j.gie.2010.04.011. Epub 2010 Jul 3. PMID 20598301